CLINICAL TRIAL: NCT02462291
Title: Effectiveness of Environmental Therapy in Patients With Alzheimer's Disease
Brief Title: New Approach for Treatment of Behavioral Disorders in Alzheimer's Disease (Alzheimer's Behavioral and Cognitive Disorders)
Acronym: ABCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Mons. Mazzali Foundation (Mantua, Italy) (Unknown)
Responsible Party: Principal Investigator, Massimo Venturelli, PhD, Research Fellow, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18201
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer Disease; Behavioral Disorders; Cognitive Impairment
Keywords: Neurological Disorders; Non Pharmacological Treatment; Ecological Therapy
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders; Cognitive Dysfunction; Nervous System Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (TR) (Experimental): A group of 80 patients with AD will perform a program of EET for 2 hours a day, 5 days a week for a total of 6 months.
  Interventions: Other: Ecological Environmental therapy
- Control group (CTRL) (No Intervention): A group of 80 patients with AD will be treated with the standard therapy.

INTERVENTIONS:
Other: Ecological Environmental therapy — The program of EET consist of the physical interaction (visual, tactile, olfactory) between natural ecological elements such as flowers, trees, grass, and the patients with AD.
  Arms: Experimental group (TR)

SUMMARY:
Alzheimer's disease (AD) is the most frequent form of dementia, causing high level of disability with elevated social costs. Alternative solutions to the standard pharmacological therapies have been studied in order to reduce the use of medications that frequently generates side effects and worsen patients' quality of life. A recent alternative treatment for AD is the Environmental Ecological Therapy (EET) that, with the use of therapeutic gardens, seems to reduce behavioral disorders (BD). However, the effectiveness of this approach is still mater of debate. Therefore, the aim of this trial will be to analyze the effects of EET, in people with severe AD.

DETAILED DESCRIPTION:
Since Homo sapiens evolved in a natural environment, an intrinsic physiologic and psychological positive reaction to nature has been developed. Accordingly, emerging literature highlights the positive effect of therapeutic gardens, as environmental ecological therapy (EET) on the reduction of behavioral disorders (BD) and the preservation of cognitive functions in patients with Alzheimer's disease (AD).

Despite these promising preliminary studies, limited data are available on the effectiveness of EET in individuals with advanced AD. Therefore, the aim of the current trial will be to evaluate the effectiveness of EET on AD symptoms in patients with advanced AD.

Participants with advanced AD will be selected from among residents of the Alzheimer's care units of the Mons. Mazzali Foundation (Mantua, Italy). Selected participants will be randomly assigned to a treatment group (TR), or to a control group (CTRL).

Participants assigned to TR group will perform a program of EET for 2 hours a day, 5 days a week for a total of 6 months. Individuals assigned to the CTRL group will be treated with a standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Person with Alzheimer's disease.

Exclusion Criteria:

* Bedridden patients.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 163 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Venturelli, Ph.D., Principal Investigator — Universita di Verona; Federico Schena, MD; Ph.D., Study Director — Universita di Verona; Nicola Smania, MD, Study Chair — Universita di Verona
Locations (1):
- Mons. Mazzali Foundation, Mantua Italy, Mantua, Italy

REFERENCES:
- [Background] Calkins MP. Evidence-based long term care design. NeuroRehabilitation. 2009;25(3):145-54. doi: 10.3233/NRE-2009-0512. PMID 19893184
- [Background] Friedrich MJ. Therapeutic environmental design aims to help patients with Alzheimer disease. JAMA. 2009 Jun 17;301(23):2430. doi: 10.1001/jama.2009.809. No abstract available. PMID 19531775
- [Background] Detweiler MB, Sharma T, Detweiler JG, Murphy PF, Lane S, Carman J, Chudhary AS, Halling MH, Kim KY. What is the evidence to support the use of therapeutic gardens for the elderly? Psychiatry Investig. 2012 Jun;9(2):100-10. doi: 10.4306/pi.2012.9.2.100. Epub 2012 May 22. PMID 22707959
- [Background] Detweiler MB, Murphy PF, Myers LC, Kim KY. Does a wander garden influence inappropriate behaviors in dementia residents? Am J Alzheimers Dis Other Demen. 2008 Feb-Mar;23(1):31-45. doi: 10.1177/1533317507309799. PMID 18276956
- [Background] Smith R, Mathews RM, Gresham M. Pre- and postoccupancy evaluation of new dementia care cottages. Am J Alzheimers Dis Other Demen. 2010 May;25(3):265-75. doi: 10.1177/1533317509357735. Epub 2010 Feb 11. PMID 20150654
- [Background] Detweiler MB, Murphy PF, Kim KY, Myers LC, Ashai A. Scheduled medications and falls in dementia patients utilizing a wander garden. Am J Alzheimers Dis Other Demen. 2009 Aug-Sep;24(4):322-32. doi: 10.1177/1533317509334036. Epub 2009 Apr 14. PMID 19366885
- [Background] Heath Y. Evaluating the effect of therapeutic gardens. Am J Alzheimers Dis Other Demen. 2004 Jul-Aug;19(4):239-42. doi: 10.1177/153331750401900410. PMID 15359562
- [Background] Rodenburg M. Special facilities for patients with Alzheimer's disease. CMAJ. 1986 Feb 15;134(4):315-6. No abstract available. PMID 3942940
- [Background] Rivasseau Jonveaux T, Batt M, Fescharek R, Benetos A, Trognon A, Bah Chuzeville S, Pop A, Jacob C, Yzoard M, Demarche L, Soulon L, Malerba G, Bouvel B. Healing gardens and cognitive behavioral units in the management of Alzheimer's disease patients: the Nancy experience. J Alzheimers Dis. 2013;34(1):325-38. doi: 10.3233/JAD-121657. PMID 23207487
- [Background] Gonzalez MT, Kirkevold M. Benefits of sensory garden and horticultural activities in dementia care: a modified scoping review. J Clin Nurs. 2014 Oct;23(19-20):2698-715. doi: 10.1111/jocn.12388. Epub 2013 Oct 15. PMID 24128125
- [Background] York SL. Residential design and outdoor area accessibility. NeuroRehabilitation. 2009;25(3):201-8. doi: 10.3233/NRE-2009-0516. PMID 19893188
- [Background] Venturelli M, Scarsini R, Muti E, Salvagno GL, Schena F. Sundowning syndrome and hypothalamic-pituitary-adrenal axis dysregulation in individuals with Alzheimer's disease: is there an association? J Am Geriatr Soc. 2013 Nov;61(11):2055-6. doi: 10.1111/jgs.12491. No abstract available. PMID 24219216
- [Background] Venturelli M, Magalini A, Scarsini R, Schena F. From Alzheimer's disease retrogenesis: a new care strategy for patients with advanced dementia. Am J Alzheimers Dis Other Demen. 2012 Nov;27(7):483-9. doi: 10.1177/1533317512459794. Epub 2012 Sep 13. PMID 22984089
- [Background] Venturelli M, Scarsini R, Schena F. Six-month walking program changes cognitive and ADL performance in patients with Alzheimer. Am J Alzheimers Dis Other Demen. 2011 Aug;26(5):381-8. doi: 10.1177/1533317511418956. Epub 2011 Aug 17. PMID 21852281
- [Background] Venturelli M, Lanza M, Muti E, Schena F. Positive effects of physical training in activity of daily living-dependent older adults. Exp Aging Res. 2010 Apr;36(2):190-205. doi: 10.1080/03610731003613771. PMID 20209421

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group (TR): A group of 82 patients with AD performed a program of EET for 2 hours a day, 5 days a week for a total of 6 months.
  Ecological Environmental therapy: The program of EET consist of the physical interaction (visual, tactile, olfactory) between natural ecological elements such as flowers, trees, grass, and the patients with AD.
- Control Group (CTRL): A group of 81 patients with AD were treated with the standard therapy.
Period: Overall Study
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Started | 82 | 81
Completed | 77 | 75
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group (TR) | Control Group (CTRL) | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (4) | 78 (5) | 77 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 121
  Male | 22 | 20 | 42
Region of Enrollment [Number; unit: participants]
  Italy | 82 | 81 | 163

OUTCOME MEASURES:

1. Primary Outcome: Evaluations of Behavioral Disorders
Description: Through the use of Neuropsychiatric Inventory (NPI), the investigators assessed the frequency and the severity of the behavioral disorders. The total scale range of the NPI is 0-144, and higher values represent worse outcome.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Scores on a scale
  PRE | 68 (19) | 66 (16)
  POST | 36 (11) | 69 (16)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 1, ANOVA; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-7.9 to 5.4]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = 33.3, 95% CI 2-sided [26.4 to 40.2]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = -31.5, 95% CI 2-sided [-38.2 to -24.8]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 1, ANOVA; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [-3.7 to 9.9]

2. Primary Outcome: Evaluation of Cognitive Status (Score 0-30)
Description: Through the use of Mini Mental State Examination (MMSE) the investigators estimated the severity and progression of cognitive impairment. MMSE is a questionnaire that examines cognitive functions including registration, attention, calculation, recall, language, ability to follow simple commands and orientation. The scale range of the MMSE tests is 0-30, and higher values represent a better outcome.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Scores on a scale
  PRE | 13.2 (1.7) | 13.1 (1.5)
  POST | 14.1 (1.6) | 12.2 (1.5)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 1, ANOVA; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = -1.94, 95% CI 2-sided [-2.6 to -1.2]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.28 to 1.61]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.52 to -0.17]

3. Secondary Outcome: Body Composition (Kilograms of Fat Free Mass)
Description: Body mass and skin-fold measurements were measured three times a day by the same experienced operator. The average value of the three measurements was calculated. Kilograms of fat free mass was estimated using a validated equation.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
kg
  PRE | 43.6 (5.9) | 42.8 (7.6)
  POST | 43.4 (6.2) | 42.1 (7.8)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.84, ANOVA; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-3.6 to 2.1]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.9, ANOVA; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-4.3 to 1.7]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.88, ANOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-3.14 to 2.69]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.89, ANOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-3.73 to 2.16]

4. Secondary Outcome: Systolic Blood Pressure (mmHg)
Description: Systolic blood pressure were measured with standard auscultatory and mercury sphygmomanometer technique.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (mmHg)
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(mmHg)
  PRE | 132 (10) | 131 (10)
  POST | 130 (9) | 132 (11)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.9, ANOVA; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-5.48 to 2.73]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.59, ANOVA; Mean Difference (Final Values) = 2.62, 95% CI 2-sided [-1.60 to 6.90]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.34, ANOVA; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-7.15 to 1.16]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.9, ANOVA; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-3.17 to 5.23]

5. Secondary Outcome: Diastolic Blood Pressure (mmHg)
Description: Diastolic blood pressure were measured with standard auscultatory and mercury sphygmomanometer technique.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (mmHg)
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(mmHg)
  PRE | 81 (5) | 81 (4)
  POST | 78 (5) | 81 (4)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.83, ANOVA; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [-1.41 to 2.14]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = 2.69, 95% CI 2-sided [0.84 to 4.53]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.010, ANOVA; Mean Difference (Final Values) = -2.14, 95% CI 2-sided [-3.94 to -0.34]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.84, ANOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-1.64 to 2.00]

6. Secondary Outcome: Blood Glucose (mg/dl)
Description: A fasted venous blood sample will be analyzed for glucose blood levels by standard techniques.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (mg/dl)
Groups:
- Control Group (CTRL): A group of 81 patients with AD was treated with the standard therapy.
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(mg/dl)
  PRE | 87.01 (3.25) | 88.41 (4.04)
  POST | 87.42 (3.76) | 88.21 (3.89)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.11, ANOVA; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-0.16 to 2.95]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.7, ANOVA; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.81 to 2.41]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.88, ANOVA; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-1.17 to 1.98]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.95, ANOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.78 to 1.39]

7. Secondary Outcome: Blood Cholesterol HDL (mg/dl)
Description: A fasted venous blood sample was analyzed for high-density lipoprotein blood levels by standard techniques.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (mg/dl)
Groups:
- Control Group (CTRL): A group of 81 patients with AD will be treated with the standard therapy.
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(mg/dl)
  PRE | 51.96 (1.19) | 51.83 (1.41)
  POST | 51.86 (1.06) | 52.29 (1.46)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.95, ANOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.67 to 0.40]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.23, ANOVA; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.12 to 0.99]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.96, ANOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.65 to 0.44]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.15, ANOVA; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.08 to 1.01]

8. Secondary Outcome: Blood Cholesterol LDL (mg/dl)
Description: A fasted venous blood sample was analyzed for low-density lipoprotein blood levels by standard techniques.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (mg/dl)
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(mg/dl)
  PRE | 98.34 (3.04) | 98.41 (2.68)
  POST | 97.86 (3.19) | 98.15 (2.69)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.84, ANOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-1.14 to 1.27]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.81, ANOVA; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.96 to 1.54]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.86, ANOVA; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.71 to 0.74]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.75, ANOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.49 to 0.97]

9. Secondary Outcome: Daily Energy Expenditure (Kcal/Day)
Description: Daily energy expenditure was measured with an Actiheart device (CamNtech, Cambridge, UK) allowing heart rate and acceleration data to be simultaneously recorded for 24 h/day for 7 consecutive days.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (Kcal/day)
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(Kcal/day)
  PRE | 1639 (134) | 1623 (155)
  POST | 1609 (128) | 1617 (154)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.94, ANOVA; Mean Difference (Final Values) = -14.7, 95% CI 2-sided [-74.4 to 44.9]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.87, ANOVA; Mean Difference (Final Values) = 8.36, 95% CI 2-sided [-53.47 to 70.20]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.78, ANOVA; Mean Difference (Final Values) = -29.70, 95% CI 2-sided [-90.19 to 30.78]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.84, ANOVA; Mean Difference (Final Values) = -6.60, 95% CI 2-sided [-67.7 to 54.5]

10. Secondary Outcome: Evaluation of Activity of Daily Life
Description: Independence and level of activities of daily life (ADL) were evaluated with the Barthel index. Levels of ADL was measured by observing each resident's daily activities (eating, bathing, grooming, dressing, transfers from bed to chair, mobility on level planes, stairs, and getting on/off the toilet). The total score of the Barthel index is 0-100, and higher values represent a better outcome.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Scores on a scale
  PRE | 51.87 (9.55) | 52.28 (9.42)
  POST | 52.49 (11.41) | 51.24 (9.40)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.74, ANOVA; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-3.73 to 4.56]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.82, ANOVA; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-5.54 to 3.04]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.59, ANOVA; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-3.57 to 4.82]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.69, ANOVA; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-5.28 to 3.19]

11. Secondary Outcome: Salivary Cortisol (Nmol/l)
Description: Levels of cortisol was measured via saliva samples using plain Sarstedt Salivette collection devices (Nümbrecht, Germany). Samples will be collected at 6.30 AM, 11.30 AM, and 6.30 PM. Immediately after collecting the saliva samples, were centrifuged for 2 min at 1,000 rpm. Purified saliva was stored in a freezer at -20 °C, and subsequently analyzed. Cortisol levels was determined by a time-resolved immunoassay with fluorometric detection.
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: (nmol/L)
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
(nmol/L)
  PRE | 10.75 (1.94) | 10.98 (2.31)
  POST | 7.82 (2.30) | 10.69 (1.71)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.9, ANOVA; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.64 to 1.09]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = 2.86, 95% CI 2-sided [1.96 to 3.76]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p < 0.01, ANOVA; Mean Difference (Final Values) = -2.92, 95% CI 2-sided [-3.80 to -2.04]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.88, ANOVA; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.17 to 0.59]

12. Secondary Outcome: Number of Medications
Time Frame: PRE and POST 6 months of treatment
Measure: Mean (Standard Deviation); unit: Number of Medications
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Number of Medications
  PRE | 3.76 (1.22) | 3.58 (1.47)
  POST | 3.10 (0.95) | 3.83 (1.57)
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Baseline; Test type: Superiority or Other; p = 0.83, ANOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.72 to 0.37]
Statistical Analysis 2: Comparison: Experimental Group (TR) vs Control Group (CTRL); After the treatment; Test type: Superiority or Other; p = 0.005, ANOVA; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [0.15 to 1.29]
Statistical Analysis 3: Comparison: Experimental Group (TR); PRE Vs POST; Test type: Superiority or Other; p = 0.013, ANOVA; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.21 to -0.09]
Statistical Analysis 4: Comparison: Control Group (CTRL); PRE Vs POST; Test type: Superiority or Other; p = 0.87, ANOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.31 to 0.81]

13. Secondary Outcome: Number of Patients Treated With Quetiapine
Time Frame: PRE and POST 6 months of treatment
Measure: Number; unit: Participants
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Participants
  PRE | 41 | 37
  POST | 35 | 37
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Test type: Superiority or Other; p = 0.910, Chi-squared; Chi-squared value = 0.542 — Power of performed test with alpha = 0.050: 0.082; 3 degrees of freedom

14. Secondary Outcome: Number of Patients Treated With Citalopram
Time Frame: PRE and POST 6 months of treatment
Measure: Number; unit: Participants
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Participants
  PRE | 55 | 57
  POST | 33 | 53
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Test type: Superiority or Other; p < 0.001, Chi-squared; Chi-squared value = 17.73 — Power of performed test with alpha = 0.050: 0.965; 3 degrees of freedom

15. Secondary Outcome: Number of Patients Treated With Donepezil
Time Frame: PRE and POST 6 months of treatment
Measure: Number; unit: Participants
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Participants
  PRE | 59 | 53
  POST | 42 | 51
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Test type: Superiority or Other; p = 0.124, Chi-squared; Chi-squared value = 5.749 — Power of performed test with alpha = 0.050: 0.488; 3 degrees of freedom

16. Secondary Outcome: Number of Patients Treated With Memantine
Time Frame: PRE and POST 6 months of treatment
Measure: Number; unit: Participants
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Participants
  PRE | 24 | 24
  POST | 23 | 22
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Test type: Superiority or Other; p = 1, Chi-squared; Chi-squared value = 0.008 — Power of performed test with alpha = 0.050: 0.050; 3 degrees of freedom

17. Secondary Outcome: Number of Patients Treated With Ticlopidin
Time Frame: PRE and POST 6 months of treatment
Measure: Number; unit: Participants
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Number analyzed (Participants) | 77 | 75
Participants
  PRE | 45 | 39
  POST | 40 | 36
Statistical Analysis 1: Comparison: Experimental Group (TR) vs Control Group (CTRL); Test type: Superiority or Other; p = 0.789, Chi-squared; Chi-squared value = 1.049 — Power of performed test with alpha = 0.050: 0.116; 3 degrees of freedom

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Experimental Group (TR): A group of 82 patients with AD will perform a program of EET for 2 hours a day, 5 days a week for a total of 6 months.
  Ecological Environmental therapy: The program of EET consist of the physical interaction (visual, tactile, olfactory) between natural ecological elements such as flowers, trees, grass, and the patients with AD.
Arm/Group | Experimental Group (TR) | Control Group (CTRL)
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No